CLINICAL TRIAL: NCT06676267
Title: Exploratory Study on the Application of Laparoscopic Surgical Systems for Gynecological and Remote Surgical Treatment.
Brief Title: Laparoscopic Surgical Systems for Gynecological and Remote Surgical Treatment.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: huaminhui
Record Dates: First submitted 2024-08-29; First posted 2024-11-06 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2024-08

CONDITIONS: Gynecological Cancer
Keywords: Laparoscopic Surgical; gynecological; Telesurgery
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- laparoscopic surgical systems (Experimental): Using the Toumai laparoscopic surgical system for gynecological surgical treatment, and combining with 5G communication technology to carry out remote surgical treatment.
  Interventions: Procedure: Laparoscopic surgery

INTERVENTIONS:
Procedure: Laparoscopic surgery — The laparoscopic surgery system is applied to gynecology and 5G remote surgical treatment.

SUMMARY:
Remote robot-assisted laparoscopic surgery will be performed for gynecological surgical treatment through 5G network, while the safety and effectiveness will be studied.

DETAILED DESCRIPTION:
This clinical study adopts a prospective, single-center, single-arm exploratory design. Remote robot-assisted laparoscopic surgery will be performed for gynecological surgical treatment through 5G network, while the safety and effectiveness will be studied.

The research process consists of three stages: the screening phase, the treatment phase and the follow-up phase. The screening phase: On the premise of meeting the inclusion and exclusion criteria, patients who voluntarily participate in robot-assisted surgery are planned to be included. Obtain written informed consent from the subjects, collect clinical data (which may include previous medical examination results), and complete relevant examinations. The treatment phase: The laparoscopic surgical system is combined with 5G network and communication technology for the surgical operation process. The follow-up phase: The physician's observational follow-up of the subjects in the study will continue up to one month post-surgery, and may be extended if necessary. During these three phases, subjects will need to undergo some medical observations or examinations to assess safety and efficacy indicators.

ELIGIBILITY:
Inclusion Criteria:

* Patients who require endoscopic surgery
* Voluntarily participate in this study and sign informed consent in writing

Exclusion Criteria:

* Patients with malignant tumors with clinical stage IV
* Those who require emergency surgery
* Presence of active bleeding, severe abnormal coagulopathy (prothrombin time (PT) or international normalized ratio (INR) greater than 1.5 times the upper limit of normal), or platelet count < 80×10^9/L
* Patient has severe cardiovascular or circulatory disease and cannot tolerate surgery
* Participated in other clinical trials in the past 1 month
* Inability to understand trial requirements, or inability to complete the study follow-up plan
* Other conditions that are considered by the investigator to be inappropriate for enrollment

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
surgical complications | From the enrollment of all subjects to one month post-surgery, assessed up to 6 months.
  The Satava classification system is used to evaluate intraoperative complications:
  Level Ⅰ: No impact on the patient, no treatment required or only conservative treatment is needed.
  Level Ⅱ: The mistake is immediately recognized and corrected, with no serious consequences.
  Level Ⅲ: The mistake is not recognized, leading to serious consequences.
  The Clavien-Dindo classification system is used to assess postoperative complications:
  Grade Ⅰ: Abnormal situations that do not require drug treatment or surgical, endoscopic, or radiologic intervention.
  Grade Ⅱ: Complications requiring drug treatment, but not requiring surgery, endoscopy, or radiologic intervention.
  Grade Ⅲ: Complications requiring surgical, endoscopic, or radiologic intervention, with Ⅲa not requiring general anesthesia and Ⅲb requiring general anesthesia.
  Grade Ⅳ: Life-threatening complications requiring ICU management, with Ⅳa for single-organ dysfunction and Ⅳb for multiple organ dysfunction.
  Grade Ⅴ: Death.

CONTACTS AND LOCATIONS:
Overall Officials: Minhui Hua, M.D., Principal Investigator — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China